CLINICAL TRIAL: NCT05742841
Title: EMERALD (Emergency Medicine Cardiovascular Risk Assessment for Lipid Disorders)
Acronym: EMERALD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00091989
Record Dates: First submitted 2023-02-15; First posted 2023-02-24 (Actual); Results first posted 2024-03-20 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2023-02

CONDITIONS: Lipid Disorder
Keywords: hyperlipidemia; cardiovascular disease; atherosclerotic cardiovascular disease
MeSH Terms: conditions — Lipid Metabolism Disorders; Hyperlipidemias; Cardiovascular Diseases; Atherosclerosis | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: 20 patients designed to assess the feasibility of Emergency Medicine Cardiovascular Risk Assessment for Lipid Disorders (EMERALD) and to explore changes in low-density lipoprotein-cholesterol (LDL-C) by initiating medical therapy in the ED
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- EMERALD protocol (Experimental): 1) ordering a lipid panel during the index ED encounter and 30-days (+/- 5 business days) after ED discharge, 2) completion of the Pooled Cohort Equations by the patient's ED provider at the index visit, and 3) starting medical therapy (moderate- or high-intensity statin/ rosuvastatin) in the ED
  Interventions: Drug: moderate- or high-intensity statin/ rosuvastatin

INTERVENTIONS:
Drug: moderate- or high-intensity statin/ rosuvastatin — moderate- or high-intensity statin (either rosuvastatin 10mg daily or rosuvastatin 40 mg daily)
  Other Names: Crestor

SUMMARY:
The EMERALD intervention involves 1) ordering an Emergency Department (ED) lipid panel, 2) calculating 10-year Atherosclerotic cardiovascular disease (ASCVD) risk using the Pooled Cohort Equations, 3) prescribing a moderate- or high-intensity statin if applicable, and 4) referring patients to outpatient care (primary care, preventive cardiology, or general cardiology, depending on risk level).

DETAILED DESCRIPTION:
EMERALD (Emergency Medicine Cardiovascular Risk Assessment for Lipid Disorders) is a pilot study seeking to determine the feasibility of initiating medical therapy for hyperlipidemia (HLD) in the Emergency Department (ED) and will collect data essential to inform a future randomized controlled trial comparing ED HLD treatment to usual care. HLD is a key cardiovascular disease (CVD) risk factor that is causally associated with atherosclerotic cardiovascular disease (ASCVD), the leading cause of US mortality and morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Department (ED) patients with chest pain
* 40-75 years old
* a low-density lipoprotein cholesterol (LDL-C) ≥70 mg/dL on an ED lipid panel or have known diabetes or Atherosclerotic Cardiovascular Disease (ASCVD)

Exclusion Criteria:

* Subject unwilling to take study medication
* Pregnancy or breastfeeding
* Inability to take study medication or, in the opinion of the Investigators/subject's doctors unsuitable for study participation
* ST-Segment Elevation Myocardial Infarction (STEMI) Activation
* ST-Segment Depression >1 mm
* On a Lipid Lowering Agent (Statin, PCSK9 Inhibitor, Bempedoic Acid, Ezetimibe, Inclisiran)
* Unstable Vitals (Blood Pressure (BP) <90, Heart Rate (HR) >120 or <50, O2 sat <90%)
* Statin Intolerance
* High-sensitivity Troponin I ≥100 ng/L
* End-Stage Renal Disease (ESRD) and/or glomerular filtration rate (GFR) <30 mL/min/1.73 m2
* Liver Cirrhosis
* Hospitalization
* Life Expectancy <1 Year
* Transfer from Another Hospital
* Prisoner
* Non-English Speaking

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Mahler, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EMERALD Protocol
Started | 22
Completed | 20
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | EMERALD Protocol
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 1
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53.5 [49.5 to 58.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Low-density Lipoprotein Cholesterol (LDL-C) Levels at Baseline and Day 30
Description: A lipid panel is a common blood test that healthcare providers use to monitor and screen for risk of cardiovascular disease. The panel includes three measurements of your cholesterol levels and a measurement of your triglycerides.
Time Frame: Baseline and Day 30
Population: only participants that qualified for study drug were analyzed - 16, not all 20 Participants
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | EMERALD Protocol
Number analyzed (Participants) | 16
mg/dL
  Baseline LDL-C | 110 [89.5 to 144.5]
  Day 30 LDL-C | 84.0 [60 to 111]
Statistical Analysis 1: Comparison: EMERALD Protocol; Test type: Superiority; Median Difference (Final Values) = -16.5

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | EMERALD Protocol
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/41/NCT05742841/Prot_003.pdf
  • Informed Consent Form (2023-06-04): https://cdn.clinicaltrials.gov/large-docs/41/NCT05742841/ICF_002.pdf